CLINICAL TRIAL: NCT07278570
Title: Magnetic Resonance Elastography to Monitor Response to Manual Therapy in Myofascial Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Ziying Yin, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-009844; 4R33AT012185-02 (NIH)
Record Dates: First submitted 2025-12-04; First posted 2025-12-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Myofascial Pain Syndrome - Lower Back; Myofascial Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tuina + Usual Care (Experimental): Participants will receive Tuina therapy twice weekly for three consecutive weeks (a total of six sessions) in addition to usual care.
  Interventions: Other: Tuina treatment; Other: Usual care
- Usual Care Only (Active Comparator): Participants will receive usual care only for three weeks, no additional manual therapy will be provided.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Tuina treatment — Tuina is a manual therapy involving techniques that apply targeted shear and stretching forces along muscular and fascial planes. Tuina therapy will be administered to subjects twice weekly for three consecutive weeks (a total of six sessions). Each session will last 30-60 minutes and will be administered by licensed Tuina practitioners trained and credentialed at Mayo Clinic.
  Arms: Tuina + Usual Care
Other: Usual care — Standard care will be followed, including a patient education course, lifestyle guidance, cognitive-behavioral therapy, and home remedies.

SUMMARY:
The purpose of this research is to develop and test new Magnetic Resonance Imaging (MRI) methods that look at how muscles and tissues under the skin (myofascial tissues) move and respond to pressure. The investigators want to see how these tissues differ between healthy people and people with pain or injury, and how they change after hands-on treatment (Tuina therapy). The results will also be compared to a group that receives standard care without Tuina therapy.

The main questions this study aims to answer are:

1. Can MR elastography (MRE) show changes in how the fascia and the layers between muscles move and stretch before and after manual therapy?
2. Do changes seen on MRE scans match changes in pain, function, and other symptoms reported by participants?
3. Can MRE measurements before treatment help predict which participants are most likely to improve with manual therapy?

In this randomized controlled trial, participants with myofascial pain will be randomly assigned (randomized) to either the Tuina group or the Usual Care group following a home-based care program without manual therapy. All treatments are noninvasive, hands-on techniques commonly used in clinical practice to reduce tissue tightness and improve movement.

Participants will be asked to undergo three MRI scans and to complete questionnaires and other standard clinical assessments about their pain, physical function, and quality of life.

DETAILED DESCRIPTION:
This research study is linked to the prior study NCT05604066 (Magnetic Resonance Elastography of Myofascial Pain Syndrome), which developed and validated the MRE techniques and biomarkers used in the current trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females (age ≥ 18 years)
* A history of chronic low back for at least 3 months. (Measured by patient history and physical exam)
* A palpable taut band or nodule within the skeletal muscle
* Hypersensitive tender spot within the taut band
* Recognition of current pain complaint by pressure on the tender nodule/taut band
* Painful limit to the full stretch range of motion

Exclusion Criteria:

* Pregnancy or breastfeeding
* Any contraindication to an MRI exam, or severe claustrophobia that would prevent safe completion of the scan
* Previous therapy in the area to be treated within 3 months
* Previous severe back injury (including fracture) or surgery
* Any neurological conditions or active systemic disease (e.g. diabetes, peripheral vascular disease, cancer, rheumatoid arthritis) that impaired sensation/pain perception
* Severe osteoarthritis
* Skin injuries in the area to be treated
* Inability to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2026-02-01 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pain, Enjoyment, and General Activity (PEG) score | Baseline, 1 day post-intervention, 3 weeks post-intervention
  The Pain, Enjoyment, and General Activity (PEG) score is a three-item questionnaire asking individuals to rate their Pain, Enjoyment of life, and General activity on a scale of 0 to 10 over the past week. The PEG score is the average of the three responses, ranging from 0 to 10, with higher scores indicating more severe pain or interference with life

CONTACTS AND LOCATIONS:
Overall Officials: Ziying Yin, Ph.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NCT05604066 - Magnetic Resonance Elastography of Myofascial Pain Syndrome — https://clinicaltrials.gov/study/NCT05604066?id=NCT05604066&rank=1